CLINICAL TRIAL: NCT05767385
Title: Fetal Cerebrovascular Autoregulation in Congenital Heart Disease and Association With Neonatal Neurobehavior
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Primary Children's Hospital (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Whitnee Hogan, MD (Assistant Professor), M.D., Assistant Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00145850; U24HL135691 (NIH)
Record Dates: First submitted 2023-03-01; First posted 2023-03-14 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Congenital Heart Disease in Children; Hypoxia; Neurodevelopmental Disorders; Complex Congenital Heart Disease
Keywords: Congenital Heart Disease; Maternal Fetal; Neonatal Neurodevelopment
MeSH Terms: conditions — Hypoxia; Neurodevelopmental Disorders; Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: Interventional Research Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Maternal Hyperoxia (MH) will be administered to pregnant patients after their standard of care fetal echocardiogram has been performed at their scheduled fetal cardiology visit at ³28 weeks gestation. The evaluation at ³28 weeks was chosen since gestational age impacts both the cardiovascular and cerebrovascular response to MH.31 The evaluation will extend the duration of the visit by approximately 30 minutes but additional evaluations or visits for the study will not be required.
  Interventions: Procedure: Single Arm; Procedure: Neonatal Neurobehavioral Scale

INTERVENTIONS:
Procedure: Single Arm — * Phase 1- Baseline: A fetal echocardiogram will be performed as part of routine standard clinical care.
  * Phase 2- MH: The participant will be placed on 8 litres of 100% FiO2 (inspired oxygen fraction) via a non-rebreather face mask for 10 minutes. After 10 minutes, additional images will be obtained. MH will be discontinued after additional imaging is complete.
  * Phase 3- Recovery: After at least 5 minutes of discontinuation of MH, additional images will be obtained to ensure any changes have returned back to baseline.
Procedure: Neonatal Neurobehavioral Scale — Neonatal Intensive Care Unit Network Neurobehavioral Scale (NNNS) evaluation: All neonates with CHD expected to undergo neonatal cardiac intervention or surgery have pre-operative NNNS assessment as PCH as standard of care. The NNNS takes approximately 30 minutes to complete. It is administered by a licensed physical, speech, or occupational therapist who has completed training and additional certification. The NNNS therapist will be blinded to the results of the fetal echocardiogram and MCA-PI.

SUMMARY:
Determine 1) the impact of abnormal fetal cerebrovascular physiology with neurodevelopmental delay (ND) outcomes and 2) how this relationship is modified by patient and environmental factors such as chronic congenital heart disease (CCHD) lesion, maternal-fetal environment, and social determinants of heath (SDOH) in a diverse population using a multicenter design.

Pregnant women will be approached during one of their fetal cardiology clinic visits.

DETAILED DESCRIPTION:
Aim 1:

Determine the association of baseline cerebrovascular resistance and reactivity and pre-operative neurobehavior in neonates with complex congenital heart disease (CCHD).

Exposures: The baseline middle cerebral artery pulsatility index (MCA-PI) and change in MCA-PI.

Analyses: Our principal analyses for Aim 1 will use separate linear regression models to relate the Neonatal Intensive Care Unit Network Neurobehavioral Scale (NNNS) attention score to 1) the baseline MCA-PI while controlling for maternal age, infant sex, race/ethnicity, and SDOH measures (maternal education, socioeconomic status (SES), insurance status), and clinical site, and 2) the change in MCA-PI adjusted for baseline MCA-PI while controlling for the same set of covariates. If the NNNS attention score distribution is skewed, we will consider transformations so that model residual plots achieve approximate normality. The covariates in the above regression analyses exclude factors that may potentially lie on the causal pathway from the MCA-PI to the attention score to avoid risk of over adjustment. In secondary analyses, 2 regression analyses will be repeated after additional adjustment for the maternal-fetal environment indicator(s), CCHD category, and age at NNNS evaluation. As a secondary analysis, we will evaluate the interaction between baseline MCA-PI and change in MCA-PI. For this analysis, we will consider dichotomizing baseline MCA-PI to facilitate interpretation of the interaction effect.

Aim 2:

Determine the impact of patient and environmental factors on cerebrovascular resistance and reactivity Exposures: Patient factors including CCHD category, indicators of the maternal-fetal environment, and SDOH

Analysis: The primary analysis for Aim 2 will investigate the joint relationship of the MCA-PI with SDOH measures and the maternal-fetal comorbidity indicator while accounting for the CCHD category (defined as Left sided obstructive lesion, Right sided obstructive lesion, Dextro-Transposition of the Great Arteries, and Other). We will apply multiple linear regression to relate the MCA-PI to the SDOH measures and a maternal-fetal comorbidity indicator for the presence of any of maternal hypertension, diabetes, pre-eclampsia, eclampsia, and abruption, prematurity, and small for gestational age. The CCHD category will also be a covariate in the regression model. Additional exploratory regression analyses will include pairwise interaction terms between the maternal-fetal comorbidity indicator(s) with the SDOH measures to assess if the association of the maternal-fetal environment indicator(s) with the MCA-PI varies across the different levels of the SDOH measures. We will perform a separate multiple regression with the change in the MCA-PI as the outcome and with the baseline MCA-PI as an additional covariate.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 18 years of age and over with a singleton fetus with known or suspected congenital heart disease anticipated to need intervention or surgery within 30 days of birth.

Exclusion Criteria:

* Known fetal chromosomal or genetic abnormalities
* Multiple gestation pregnancy
* Fetal extra-cardiac anomalies

Ages: 0 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Pregnant females with fetus diagnosis congenital heart disease.
Enrollment: 150 (Estimated)
Dates: Start 2021-12-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pre-operative Neonatal Network Neurobehavioral Scale (NNNS) attention scores | <=30 days of life
  The NeoNatal Neurobehavioral Scale (NNNS-II) examines the neurobehavioral organization, neurological reflexes, motor development - active and passive tone, and signs of stress and withdrawal of the at-risk and drug-exposed infant
Baseline MCA-PI and change in MCA-PI with Maternal Hyperoxia | <= 30 days of life
  The fetal middle cerebral artery (MCA) pulsatility index (PI)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of California San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Maine Medical Center, Scarborough, Maine
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marino BS, Lipkin PH, Newburger JW, Peacock G, Gerdes M, Gaynor JW, Mussatto KA, Uzark K, Goldberg CS, Johnson WH Jr, Li J, Smith SE, Bellinger DC, Mahle WT; American Heart Association Congenital Heart Defects Committee, Council on Cardiovascular Disease in the Young, Council on Cardiovascular Nursing, and Stroke Council. Neurodevelopmental outcomes in children with congenital heart disease: evaluation and management: a scientific statement from the American Heart Association. Circulation. 2012 Aug 28;126(9):1143-72. doi: 10.1161/CIR.0b013e318265ee8a. Epub 2012 Jul 30. PMID 22851541
- [Background] Donofrio MT, Duplessis AJ, Limperopoulos C. Impact of congenital heart disease on fetal brain development and injury. Curr Opin Pediatr. 2011 Oct;23(5):502-11. doi: 10.1097/MOP.0b013e32834aa583. PMID 21881507
- [Background] McQuillen PS, Miller SP. Congenital heart disease and brain development. Ann N Y Acad Sci. 2010 Jan;1184:68-86. doi: 10.1111/j.1749-6632.2009.05116.x. PMID 20146691
- [Background] Limperopoulos C, Tworetzky W, McElhinney DB, Newburger JW, Brown DW, Robertson RL Jr, Guizard N, McGrath E, Geva J, Annese D, Dunbar-Masterson C, Trainor B, Laussen PC, du Plessis AJ. Brain volume and metabolism in fetuses with congenital heart disease: evaluation with quantitative magnetic resonance imaging and spectroscopy. Circulation. 2010 Jan 5;121(1):26-33. doi: 10.1161/CIRCULATIONAHA.109.865568. Epub 2009 Dec 21. PMID 20026783
- [Background] Peyvandi S, Xu D, Wang Y, Hogan W, Moon-Grady A, Barkovich AJ, Glenn O, McQuillen P, Liu J. Fetal Cerebral Oxygenation Is Impaired in Congenital Heart Disease and Shows Variable Response to Maternal Hyperoxia. J Am Heart Assoc. 2021 Jan 5;10(1):e018777. doi: 10.1161/JAHA.120.018777. Epub 2020 Dec 21. PMID 33345557
- [Background] Dimitropoulos A, McQuillen PS, Sethi V, Moosa A, Chau V, Xu D, Brant R, Azakie A, Campbell A, Barkovich AJ, Poskitt KJ, Miller SP. Brain injury and development in newborns with critical congenital heart disease. Neurology. 2013 Jul 16;81(3):241-8. doi: 10.1212/WNL.0b013e31829bfdcf. Epub 2013 Jun 14. PMID 23771484
- [Background] Vesoulis ZA, Mathur AM. Cerebral Autoregulation, Brain Injury, and the Transitioning Premature Infant. Front Pediatr. 2017 Apr 3;5:64. doi: 10.3389/fped.2017.00064. eCollection 2017. PMID 28421173
- [Background] Oros D, Figueras F, Cruz-Martinez R, Padilla N, Meler E, Hernandez-Andrade E, Gratacos E. Middle versus anterior cerebral artery Doppler for the prediction of perinatal outcome and neonatal neurobehavior in term small-for-gestational-age fetuses with normal umbilical artery Doppler. Ultrasound Obstet Gynecol. 2010 Apr;35(4):456-61. doi: 10.1002/uog.7588. PMID 20178115
- [Background] Hogan WJ, Moon-Grady AJ, Zhao Y, Cresalia NM, Nawaytou H, Quezada E, Brook M, McQuillen P, Peyvandi S. Fetal cerebrovascular response to maternal hyperoxygenation in congenital heart disease: effect of cardiac physiology. Ultrasound Obstet Gynecol. 2021 May;57(5):769-775. doi: 10.1002/uog.22024. Epub 2021 Apr 13. PMID 32202689
- [Background] Donofrio MT, Bremer YA, Schieken RM, Gennings C, Morton LD, Eidem BW, Cetta F, Falkensammer CB, Huhta JC, Kleinman CS. Autoregulation of cerebral blood flow in fetuses with congenital heart disease: the brain sparing effect. Pediatr Cardiol. 2003 Sep-Oct;24(5):436-43. doi: 10.1007/s00246-002-0404-0. PMID 14627309
- [Background] Williams IA, Tarullo AR, Grieve PG, Wilpers A, Vignola EF, Myers MM, Fifer WP. Fetal cerebrovascular resistance and neonatal EEG predict 18-month neurodevelopmental outcome in infants with congenital heart disease. Ultrasound Obstet Gynecol. 2012 Sep;40(3):304-9. doi: 10.1002/uog.11144. Epub 2012 Aug 2. PMID 22351034
- [Background] Hahn E, Szwast A, Cnota J 2nd, Levine JC, Fifer CG, Jaeggi E, Andrews H, Williams IA. Association between fetal growth, cerebral blood flow and neurodevelopmental outcome in univentricular fetuses. Ultrasound Obstet Gynecol. 2016 Apr;47(4):460-5. doi: 10.1002/uog.14881. Epub 2016 Feb 18. PMID 25900850
- [Background] Szwast A, Putt M, Gaynor JW, Licht DJ, Rychik J. Cerebrovascular response to maternal hyperoxygenation in fetuses with hypoplastic left heart syndrome depends on gestational age and baseline cerebrovascular resistance. Ultrasound Obstet Gynecol. 2018 Oct;52(4):473-478. doi: 10.1002/uog.18919. Epub 2018 Sep 3. PMID 28976608
- [Background] Sanapo L, Al-Shargabi T, Ahmadzia HK, Schidlow DN, Donofrio MT, Hitchings L, Khoury A, Larry Maxwell G, Baker R, Bulas DI, Gomez LM, du Plessis AJ. Fetal acute cerebral vasoreactivity to maternal hyperoxia in low-risk pregnancies: a cross-sectional study. Prenat Diagn. 2020 Jun;40(7):813-824. doi: 10.1002/pd.5694. Epub 2020 Apr 20. PMID 32274806
- [Background] Rasanen J, Wood DC, Debbs RH, Cohen J, Weiner S, Huhta JC. Reactivity of the human fetal pulmonary circulation to maternal hyperoxygenation increases during the second half of pregnancy: a randomized study. Circulation. 1998 Jan 27;97(3):257-62. doi: 10.1161/01.cir.97.3.257. PMID 9462527
- [Background] Hogan WJ, Winter S, Pinto NM, Weng C, Sheng X, Conradt E, Wood J, Puchalski MD, Tani LY, Miller TA. Neurobehavioral evaluation of neonates with congenital heart disease: a cohort study. Dev Med Child Neurol. 2018 Dec;60(12):1225-1231. doi: 10.1111/dmcn.13912. Epub 2018 May 10. PMID 29748956
- [Background] Gakenheimer-Smith L, Glotzbach K, Ou Z, Presson AP, Puchalski M, Jones C, Lambert L, Delgado-Corcoran C, Eckhauser A, Miller T. The Impact of Neurobehavior on Feeding Outcomes in Neonates with Congenital Heart Disease. J Pediatr. 2019 Nov;214:71-78.e2. doi: 10.1016/j.jpeds.2019.06.047. Epub 2019 Aug 8. PMID 31402138
- [Background] Ebbing C, Rasmussen S, Kiserud T. Middle cerebral artery blood flow velocities and pulsatility index and the cerebroplacental pulsatility ratio: longitudinal reference ranges and terms for serial measurements. Ultrasound Obstet Gynecol. 2007 Sep;30(3):287-96. doi: 10.1002/uog.4088. PMID 17721916
- [Background] Williams IA, Fifer C, Jaeggi E, Levine JC, Michelfelder EC, Szwast AL. The association of fetal cerebrovascular resistance with early neurodevelopment in single ventricle congenital heart disease. Am Heart J. 2013 Apr;165(4):544-550.e1. doi: 10.1016/j.ahj.2012.11.013. Epub 2013 Feb 13. PMID 23537971